CLINICAL TRIAL: NCT06249581
Title: Pharmacokinetics of Nicorandil 40 mg Extended-Release Capsules: A Single-Dose, Open-Label, Randomized, Two-Sequence, Two-Treatment, Two-Period Crossover Study in Healthy Subjects Under Fasting and Fed Conditions
Brief Title: Pharmacokinetics of AUX-001 40mg Once-daily in Healthy Subjects Under Fasting and Fed Conditions
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Auxilius Pharma sp.z.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-506085-31-00
Record Dates: First submitted 2023-12-20; First posted 2024-02-08 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Chronic Stable Angina
Keywords: Pharmacokinetics; Bioavailability; Safety; Tolerability; Fasting; Fed
MeSH Terms: conditions — Angina, Stable; Fasting; Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Intervention Model Description: Single-dose clinical trial with healthy volunteers sequentially using a single dose of AUX-001 under fasting and thereafter under fed conditions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: fasting (Experimental): AUX-001 40mg QD
  Interventions: Drug: AUX-001 40mg once-daily
- Arm B: fed (Experimental): AUX-001 40mg QD
  Interventions: Drug: AUX-001 40mg once-daily

INTERVENTIONS:
Drug: AUX-001 40mg once-daily — AUX-001 (extended-release nicorandil) 40mg QD (once-daily)
  Other Names: Food effect

SUMMARY:
Exploratory, single-dose, open-label, pharmacokinetic study to establish uptake, plasma levels safety and tolerability of orally administered AUX-001 on an empty stomach (i.e, fasting) as well as after a meal (i.e. fed) in healthy volunteers.

DETAILED DESCRIPTION:
This is a first-in-human, exploratory, single-dose, open-label pharmacokinetic study to explore the uptake, and systemic distribution of orally administered AUX-001 in healthy volunteers on an empty stomach (i.e, fasting) as well as after a meal (i.e. fed) in male and female healthy volunteers age 18 to 55 to establish pharmacokinetics, safety, tolerability and whether the medication can be given independent of any food effect.

ELIGIBILITY:
Inclusion Criteria:

1. Free written informed consent signed and dated prior to any procedure required by the study.
2. Male or female subject between 18 and 55years, inclusive, at the time of signing the informed consent.
3. Body mass index (BMI) of 18.0 to 31.0 kg/m2, inclusive.
4. No clinically relevant diseases captured in medical history.
5. No clinically relevant abnormalities on physical examination.
6. No clinically relevant abnormalities on vital signs.
7. No clinically relevant abnormalities on 12-lead EKG.
8. No clinically relevant abnormalities on laboratory tests.
9. Neg. test results on anti-HIV-1Ab and anti-HIV-2Ab, HbsAG and anti-HCVAb
10. Non-smoker or ex-smoker
11. Willingness to accept and comply with all study procedures and restrictions.
12. Female subject of a) non-child-bearing potential or b) of childbearing potential and agrees to use an accepted, highly effective contraceptive method until the end of the study.

Exclusion Criteria:

1. Known hypersensitivity/allergy reaction to the study drug substance or any of the excipients.
2. Known severe hypersensitivity reaction to any other drug.
3. Any medical condition (e.g., gastrointestinal, renal or hepatic, including peptic ulcer, inflammatory bowel disease or pancreatitis) or surgical condition (e.g., cholecystectomy, gastrectomy) that may affect drug pharmacokinetics (absorption, distribution, metabolism or excretion) or subject's safety.
4. History of glucose-6-phosphate dehydrogenase deficiency.
5. History of severe hypotension or shock.
6. History of acute pulmonary edema, heart failure, coronary artery disease or myocardial infarction.
7. History of orthostatic hypotension, collapse, fainting, syncope, or vasovagal reaction.
8. History of substance or alcohol abuse within the previous 2 years.
9. Use of contact lenses.
10. SBP <95 mmHg and/or DBP <45 mmHg.
11. Serum transaminases alanine aminotransferase (ALT) or aspartate aminotransferase (AST) above the upper limit of the normal range.
12. Estimated renal creatinine clearance (CLCr) below the lower limit of normal range, based on creatinine clearance calculation by the Cockcroft-Gault formula and normalized to an average body surface area of 1.73 m2.
13. Positive result in drugs-of-abuse or ethanol tests.
14. Use of a depot injection or an implant of any drug (except for contraceptives) within the previous 6 months.
15. Average weekly alcohol consumption of >14 units for males and >7 units for females within the previous 6 months.
16. Average daily consumption of methylxanthines-containing beverages or food (e.g., coffee, tea, cola, sodas, chocolate) equivalent to >500 mg of methylxanthines.
17. Participation in any clinical trial within the previous 2 months.
18. Participation in more than 2 clinical trials within the previous 12 months.
19. Blood donation or significant blood loss (≥ 450 mL) due to any reason or had plasmapheresis within the previous 2 months.
20. Difficulty in fasting or any dietary restriction such as lactose intolerance, vegan, low-fat, low sodium, etc., that may interfere with the diet served during the study.
21. Veins unsuitable for intravenous puncture on either arm.
22. Difficulty in swallowing capsules or tablets.
23. If woman of childbearing potential (WOCBP), positive pregnancy test.
24. If woman, she is breast-feeding.
25. Any other condition that the Investigator considers to render the subject unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-02-08 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Area under the curve over 24 hours [AUC0-24h)] of nicorandil under fasting conditions | 24 hours
  Total nicorandil plasma concentration over 24 hours under fasting conditions
Area under the curve over 24 hours [AUC0-24h)] of nicorandil under fed conditions | 24 hours
  Total nicorandil plasma concentration over 24 hours under fed conditions
Maximum Plasma Concentration [Cmax] of nicorandil under fasting conditions | 24 hours
  Peak plasma concentration under fasting conditions in mcg/ml
Maximum Plasma Concentration [Cmax] of nicorandil under fed conditions | 24 hours
  Peak plasma concentration under fed conditions in mcg/ml
24 hour Area Under the Curve [AUC0-24h] of N-(2-hydroxyethyl) nicotinamide under fasting conditions | 24 hours
  24 hour Total Plasma Concentration of nicorandil's main metabolite under fasting conditions
24h hour Area Under the Curve [AUC0-24h] of N-(2-hydroxyethyl) nicotinamide under fed conditions | 24 hours
  Total Plasma Concentration of nicorandil's main metabolite under fed conditions

SECONDARY OUTCOMES:
Treatment-emergent adverse events [TEAE] under fasting conditions | 24 hours
  Occurrence of treatment-emergent adverse events (TEAEs) including vital signs, pulse oximetry, EKG, liver function tests [LFT] under fasting conditions
Treatment-emergent adverse events [TEAE] under fed conditions | 24 hours
  Occurrence of treatment-emergent adverse events (TEAEs) including vital signs, pulse oximetry, EKG, liver function tests [LFT] under fed conditions

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fonseca, MD, Principal Investigator — Blueclinical, Ltd.; Uwe P Tigör, MD, Study Director — Auxilius Pharma
Locations (1):
- BlueClinical, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No